CLINICAL TRIAL: NCT04188184
Title: Topical Use of Tranexamic Acid Versus Epinephrine to Optimize Surgical Field During Exploratory Tympanotomy
Brief Title: Tranexamic Acid Versus Epinephrine During Exploratory Tympanotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, Director, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17300198
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexmic acid (Active Comparator): received topical 1 gram of TXA diluted in 200 ml of normal saline (0.9%) for topical use to rinse the bleeding sites and soak the used gauze for local compression.
  Interventions: Drug: Tranexamic Acid
- Epinephrine roup (Active Comparator): received Epinephrine 1 mg diluted in 200 ml normal saline (0.9%) for topical use to rinse the bleeding sites and soak the used gauze for local compression.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Tranexamic Acid — received topical 1 gram of TXA diluted in 200 ml of normal saline (0.9%) for topical use to rinse the bleeding sites and soak the used gauze for local compression.
  Arms: tranexmic acid
Drug: Epinephrine — received Epinephrine 1 mg diluted in 200 ml normal saline (0.9%) for topical use to rinse the bleeding sites and soak the used gauze for local compression.
  Arms: Epinephrine roup

SUMMARY:
Exploratory tympanotomy is surgical access to the middle ear, made for diagnosis and management of unexplained conductive hearing loss, performed under an oto-microscope across the external auditory canal after tympanic membrane elevation to explore the middle ear structures

DETAILED DESCRIPTION:
Epinephrine is a vasoconstrictor searched intensively for ptimization of the surgical field during microscopic ear and sinus surgeries with controversial results given the possible cardiovascular complication in case of systemic absorption,especially in vulnerable cardiac patients.Tranexamic acid (TXA) as an antifibrinolytic medication is used to treat or prevent excessive bleeding in significant trauma, surgery, tooth removal, or nasal bleeding, discovered by Japanese researchers. TXA, given either oral or intravenous, is a derivative of lysine amino acid; it acts reversibly on the lysine binding sites to block it on the plasminogen molecules. TXA consequently hinders the stimulation of plasminogen competitively, thus reduces its conversion into plasmin. Plasminogen is the enzyme that leads to the degradation of a fibrin clot, fibrinogen, and other plasma proteins, such as factors V and VIII. More than 95% of TXA intravenous administered dose eliminated unchanged through the urinary system. Twenty-four hours after intravenous administration of TXA has demonstrated accumulative excretion of approximately 90%, whereas only 3% is bound to plasminogen. TXA is minimally excreted in breast milk while it can freely cross the blood brain barrier and the placenta .

ELIGIBILITY:
Inclusion Criteria:

* 18 - 60 years old
* ASA (I and II)
* Hb level > 10 mg/dl
* elective ear exploratory tympanotomy surgery under general anesthesia.

Exclusion Criteria:

* Allergy to TXA
* bleeding/coagulation disorders
* psychiatric illness
* acute and chronic renal failure
* heparin use within 48 hrs or aspirin use within seven days before surgery,
* pregnancy
* liver cirrhosis
* color blindness
* cardiac stent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
State of surgical field categorized by surgeons based on Boezaart classification | 2 hour
  Grade Description 0 No bleeding (cadaveric conditions)
  1. Slight bleeding: no suctioning required
  2. Slight bleeding: occasional suctioning required
  3. Slight bleeding: frequent suctioning required, bleeding threatens surgical field a few seconds after suction is removed
  4. Moderate bleeding: frequent suctioning required and bleeding threatens surgical field directly after suction is removed
  5. Severe bleeding: constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible

SECONDARY OUTCOMES:
bleeding volume | 2 hour
  The quantity of blood (ml) = (mass of used + fresh gauze - weight of all sponges before surgery) / 1.05.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut university, Asyut
  - Faculty of Medicine, Asyut